CLINICAL TRIAL: NCT02120443
Title: ivWatch Model 400: Device Validation for Non-Infiltrated Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Principal Investigator, Garret Bonnema, Chief Science Officer, ivWatch, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVW400CS-05
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Infiltration of Peripheral IV Therapy
Keywords: infiltration; extravasation; peripheral intravenous therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-Infiltrated Tissue (Experimental): The ivWatch Model 400 monitored a common peripheral IV site over a 24 hour observation period.
  Interventions: Device: ivWatch Model 400

INTERVENTIONS:
Device: ivWatch Model 400 — The ivWatch Model 400 monitored tissue at common IV sites over a 24 hour period.

SUMMARY:
A single arm study of 40 adult volunteers to assess the safety and efficacy of the ivWatch Model 400 when observing non-infiltrated (normal) tissues at common peripheral IV therapy sites.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Pass health screen
* 18 years or older

Exclusion Criteria:

* Fail health screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ivWatch, LLC, Williamsburg, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Infiltrated Tissue
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Non-Infiltrated Tissue
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (13.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 43
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (5.4)
Skin Pigmentation [Mean (Standard Deviation); unit: units on a scale] — Skin pigmentation was scored from 1 to 3 where 1 represents light skin pigmentation, 2 represents medium skin pigmentation, and 3 represents dark skin pigmentation.
  units on a scale | 1.84 (0.84)

OUTCOME MEASURES:

1. Primary Outcome: Normal Tissue Red Notification Rate
Description: The ivWatch Model 400 issues red notifications to communicate the need for a clinician to check an IV site. A red notification suggests an increased likelihood that an IV infiltration may be occurring, with a greater likelihood relative to a yellow notification. This measure describes the average number of red notifications issued by the ivWatch device in a given day when monitoring normal, non-infiltrated tissues. The 95% confidence interval for the red notification rate was calculated using the Clopper-Pearson method.
Time Frame: 24 hours
Population: Three subjects were excluded from analysis due to significant protocol deviations.
Measure: Mean (95% Confidence Interval); unit: red notifications per day
Arm/Group | Non-Infiltrated Tissue
Number analyzed (Participants) | 40
red notifications per day | 0.24 [0.11 to 0.45]

2. Secondary Outcome: Normal Tissue Yellow Notification Rate
Description: The ivWatch Model 400 issues yellow notifications to communicate the need for a clinician to check an IV site. A yellow notification suggests an increased likelihood that an IV infiltration may be occurring, although at a lower likelihood relative to a red notification. This measure describes the average number of yellow notifications issued by the ivWatch device in a given day when monitoring normal, non-infiltrated tissues. The 95% confidence interval for the yellow notification rate was calculated using the Clopper-Pearson method.
Time Frame: 24 hours
Population: Three participants were excluded due to significant protocol deviations.
Measure: Mean (95% Confidence Interval); unit: yellow notifications per day
Arm/Group | Non-Infiltrated Tissue
Number analyzed (Participants) | 40
yellow notifications per day | 0.51 [0.31 to 0.79]

3. Secondary Outcome: Significant Skin Irritation or Disruption to Skin Integrity
Description: The number of IV sites with significant skin irritation or disruption to skin integrity assessed at the end of the study. The Clopper-Pearson method was used for estimating the binomial proportion confidence interval.
Time Frame: 24 hours
Population: Three participants were excluded for significant protocol deviations.
Measure: Number (95% Confidence Interval); unit: IV sites
Arm/Group | Non-Infiltrated Tissue
Number analyzed (Participants) | 40
IV sites | 0 [0 to 0.0881]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the individual studies (approximately 24 hours)
Arm/Group | Non-Infiltrated Tissue
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes